CLINICAL TRIAL: NCT03560531
Title: A Phase 1/2 Open Label, Multicenter Study to Assess the Safety, Tolerability, Pharmacokinetics, and Anti-Tumor Activity of ZN-c5 Alone and in Combination With Palbociclib in Subjects With Estrogen-Receptor Positive, Human Epidermal Growth Factor Receptor-2 Negative Advanced Breast Cancer
Brief Title: A Study of ZN-c5 in Subjects With Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Zeno Alpha Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZN-c5-001
Record Dates: First submitted 2018-06-05; First posted 2018-06-18 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Breast Cancer
Keywords: Estrogen receptor; Hormone receptor; Selective estrogen receptor degrader; Hormone sensitive; Phase 1 Dose Escalation; Phase 2 Combination; Phase 1 Dose Expansion; Phase 2 Monotherapy
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Intervention Model Description: Dose escalation cohorts are planned in monotherapy and combination as well as monotherapy dose expansion, and monotherapy and combination Phase 2.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZN-c5 monotherapy (Experimental): Dose escalation cohorts are planned to determine maximum tolerated dose(MTD) or recommended phase 2 dose (RP2D) of ZN-c5 as well as expansion cohorts and a Phase 2 cohort.
  Interventions: Drug: ZN-c5
- ZN-c5 + palbociclib combination therapy (Experimental): Dose escalation cohorts are planned to determine maximum tolerated dose(MTD) or recommended phase 2 dose (RP2D) of ZN-c5 in combination with palbociclib as well as a Phase 2 cohort.
  Interventions: Drug: ZN-c5; Drug: Palbociclib

INTERVENTIONS:
Drug: ZN-c5 — ZN-c5 is a study drug
Drug: Palbociclib — Palbociclib (IBRANCE®) is an approved drug
  Other Names: IBRANCE®
  Arms: ZN-c5 + palbociclib combination therapy

SUMMARY:
This is a Phase 1/2, open-label, multicenter, dose-escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of ZN-c5 administered orally in subjects with advanced estrogen receptor positive, human epidermal growth factor receptor 2 negative (ER+/HER2-) breast cancer. ZN-c5 will be evaluated both as monotherapy and in combination with palbociclib (IBRANCE®).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years of age

  * Women can be postmenopausal, as defined by at least one of the following:
  * Age ≥ 60 years;
  * Age < 60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and serum estradiol and follicle-stimulating hormone level within the laboratory's reference range for postmenopausal females;
  * Documented bilateral oophorectomy; or can be peri- or premenopausal, however, they must receive a gonadotrophin-releasing hormone agonist beginning at least 4 weeks prior to the first dose of study medication.
* Histologically or cytologically confirmed diagnosis of advanced (metastatic or locoregionally recurrent) adenocarcinoma of the breast, not amenable to any potential curative intervention
* Estrogen Receptor (ER) positive disease
* Human Epidermal Growth Factor Receptor 2 (HER2) negative disease
* Documented prior response to endocrine therapy for metastatic disease (stable disease, partial response, or complete response by RECIST v1.1 criteria) lasting > 6 months
* Evaluable or measurable disease by RECIST v1.1. Tumor lesions previously irradiated or subjected to other locoregional therapy will only be deemed measurable if progression at the treated site after completion of therapy is clearly documented.

Exclusion Criteria:

* Prior anticancer or investigational drugs for the treatment of ER+/HER2 negative advanced breast cancer within the following windows:

  * Tamoxifen, aromatase inhibitor, fulvestrant, or other anti-cancer endocrine therapy < 14 days before first dose of study treatment
  * Any chemotherapy < 28 days before first dose of study, except for Phase 2 monotherapy which requires no prior chemotherapy treatment.
  * Any investigational drug therapy < 28 days or 5 half-lives (whichever is shorter) prior to first dose of study treatment
* Unexplained symptomatic endometrial disorders (including, but not limited to endometrial hyperplasia, dysfunctional uterine bleeding, or cysts)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2022-04-26 (Actual); Study Completion 2022-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeno Alpha, Inc., Study Director — Zeno Alpha Inc.
Locations (38):
- United States (11):
  - Site 3, Tucson, Arizona
  - Site 5, Los Angeles, California
  - Site 48, Bethesda, Maryland
  - Site 47, St Louis, Missouri
  - Site 7, New York, New York
  - Site 2, New York, New York
  - Site 50, Charleston, South Carolina
  - Site 4, Nashville, Tennessee
  - Site 1, Houston, Texas
  - Site 8, Houston, Texas
  - Site 6, Seattle, Washington
- Belarus (2):
  - Site 46, Minsk
  - Site 45, Vitebsk
- Bosnia and Herzegovina (3):
  - Site 10, Banja Luka
  - Site 9, Sarajevo
  - Site 11, Tuzla
- Czechia (3):
  - Site 29, Brno
  - Site 28, Olomouc
  - Site 30, Prague
- Hungary (3):
  - Site 51, Budapest
  - Site 35, Kecskemét
  - Site 37, Pécs
- Lithuania (2):
  - Site 17, Kaunas
  - Site 16, Vilnius
- Russia (5):
  - Site 40, Nizhny Novgorod
  - Site 52, Omsk
  - Site 41, Pyatigorsk
  - Site 39, Saint Petersburg
  - Site 42, Yekaterinburg
- Serbia (4):
  - Site 18, Belgrade
  - Site 19, Belgrade
  - Site 21, Niš
  - Site 20, Novi Sad
- Ukraine (5):
  - Site 25, Cherkasy
  - Site 27, Kharkiv
  - Site 24, Kropyvnytskyi
  - Site 26, Kryvyi Rih
  - Site 23, Kyiv

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was initiated on 30 November 2018 and completed on 22 December 2022 (last participant last visit). 29 centers in Belarus, Bosnia and Herzegovina, the Czech Republic, Hungary, Lithuania, Russia, Serbia, Ukraine, and the United States enrolled the participants.
Groups:
- Phase 1 (Monotherapy): ZN-c5 50 mg QD: Participants who received ZN-c5 50 mg once daily (QD) in Phase 1 were included in this arm.
- Phase 1 (Monotherapy): ZN-c5 75 mg QD: Participants who received ZN-c5 75 mg QD in Phase 1 were included in this arm.
- Phase 1 (Monotherapy): ZN-c5 100 mg QD: Participants who received ZN-c5 100 mg QD in Phase 1 were included in this arm.
- Phase 1 (Monotherapy): ZN-c5 75 mg BID: Participants who received ZN-c5 75 mg twice daily (BID) in Phase 1 were included in this arm.
- Phase 1 (Monotherapy): ZN-c5 150 mg QD: Participants who received ZN-c5 150 mg QD in Phase 1 were included in this arm.
- Phase 1 (Monotherapy): ZN-c5 150 mg BID: Participants who received ZN-c5 150 mg BID in Phase 1 were included in this arm.
- Phase 1 (Monotherapy): ZN-c5 300 mg QD: Participants who received ZN-c5 300 mg QD in Phase 1 were included in this arm.
- Phase 2 (Monotherapy): ZN-c5 50 mg QD: Participants who received ZN-c5 50 mg QD in Phase 2 were included in this arm.
- Phase 1 (Combination Therapy): ZN-c5 25mg QD + Palbociclib: Participants who received ZN-c5 25 mg QD along with Palbociclib (IBRANCE®) in Phase 1 were included in this arm.
- Phase 1 (Combination Therapy): ZN-c5 25mg BID + Palbociclib: Participants who received ZN-c5 25 mg BID along with Palbociclib (IBRANCE®) in Phase 1 were included in this arm.
- Phase 1 (Combination Therapy): ZN-c5 50mg QD + Palbociclib: Participants who received ZN-c5 50 mg QD along with Palbociclib (IBRANCE®) in Phase 1 were included in this arm.
- Phase 1 (Combination Therapy): ZN-c5 50mg BID + Palbociclib: Participants who received ZN-c5 50 mg BID along with Palbociclib (IBRANCE®) in Phase 1 were included in this arm.
- Phase 1 (Combination Therapy): ZN-c5 100mg QD + Palbociclib: Participants who received ZN-c5 100 mg QD along with Palbociclib (IBRANCE®) in Phase 1 were included in this arm.
- Phase 1 (Combination Therapy): ZN-c5 150mg QD + Palbociclib: Participants who received ZN-c5 150 mg QD along with Palbociclib (IBRANCE®) in Phase 1 were included in this arm.
Period: Overall Study
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Combination Therapy): ZN-c5 25mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 25mg BID + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 50mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 50mg BID + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 100mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 150mg QD + Palbociclib
Started | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75 | 10 | 5 | 18 | 2 | 12 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75 | 10 | 5 | 18 | 2 | 12 | 3
Not completed — Death | 4 | 1 | 1 | 2 | 6 | 1 | 4 | 8 | 1 | 3 | 2 | 0 | 4 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 0 | 0 | 2 | 0
Not completed — Study end per-protocol | 1 | 1 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Early study termination by sponsor | 9 | 0 | 0 | 4 | 8 | 2 | 5 | 64 | 7 | 2 | 16 | 2 | 6 | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set consisted of all participants who received ≥1 dose of study drug and was used in the analyses of participant characteristics and efficacy endpoints.
Groups:
- Phase 1 (Monotherapy): ZN-c5 50 mg QD: Participants who received ZN-c5 50 mg QD in Phase 1 were included in this arm.
- Phase 1 (Monotherapy): ZN-c5 75 mg BID: Participants who received ZN-c5 75 mg BID in Phase 1 were included in this arm.
- Total: Total of all reporting groups
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Combination Therapy): ZN-c5 25mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 25mg BID + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 50mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 50mg BID + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 100mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 150mg QD + Palbociclib | Total
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75 | 10 | 5 | 18 | 2 | 12 | 3 | 181
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 11 | 3 | 3 | 3 | 10 | 2 | 5 | 39 | 6 | 3 | 8 | 2 | 8 | 2 | 105
  >=65 years | 5 | 0 | 0 | 3 | 5 | 1 | 5 | 36 | 4 | 2 | 10 | 0 | 4 | 1 | 76
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75 | 10 | 5 | 18 | 2 | 11 | 3 | 180
  Male | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
  Black or African American | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
  White | 12 | 3 | 3 | 5 | 12 | 3 | 9 | 74 | 8 | 5 | 17 | 1 | 10 | 3 | 165
  Not Reported | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 6
  Other | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 3 | 3 | 6 | 15 | 3 | 8 | 13 | 10 | 5 | 18 | 2 | 12 | 3 | 109
  Europe | 8 | 0 | 0 | 0 | 0 | 0 | 2 | 62 | 0 | 0 | 0 | 0 | 0 | 0 | 72

OUTCOME MEASURES:

1. Primary Outcome: Clinical Benefit Rate (CBR) for ZN-c5 as a Monotherapy
Description: CBR is defined as the number of participants who have at least 1 confirmed response of complete response (CR) or partial response (PR) (only if participant has measurable disease), or stable disease (SD) >= 24 weeks (or non-CR/non-progressive disease (PD) >=24 weeks for participants with non-measurable disease) prior to any evidence of progression.
Time Frame: 24 weeks
Population: Full Analysis Set consisted of all participants who received >=1 dose of study drug and was used in the analyses of participant characteristics and efficacy endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
Participants | 7 | 0 | 1 | 1 | 4 | 1 | 5 | 38

2. Primary Outcome: Best Overall Response (BOR) for ZN-c5 as a Monotherapy
Description: Best overall response was summarized categorically based on the four RECIST categories: CR, PR, SD and PD.
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  PR | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3
  SD | 13 | 1 | 1 | 6 | 10 | 3 | 7 | 50
  SD ≥24 weeks | 7 | 0 | 1 | 1 | 3 | 1 | 4 | 35
  8 weeks < SD <24 weeks | 6 | 1 | 0 | 5 | 7 | 2 | 3 | 15
  PD | 3 | 2 | 2 | 0 | 4 | 0 | 1 | 19
  Non-Responders (NR) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Not Evaluable (NE) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Monotherapy Only: Percentage of Participants With Progression-Free Survival (PFS) at 2 Months
Description: PFS is defined as the time (in months) from the date of first dosing until the date of objective PD (as defined by RECIST version 1.1) or death (by any cause in the absence of progression), whichever occurs earlier. Kaplan-Meier estimates at 2 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 2 months
Population: The Tumor Response-Evaluable Set includes all participants in the full analysis set with at least 1 evaluable postbaseline response assessment using RECIST 1.1.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 9 | 72
percentage of participants | 87.1 [57.3 to 96.6] | 66.7 [5.4 to 94.5] | 33.3 [0.9 to 77.4] | 100.0 [100.0 to 100.0] | 73.3 [43.6 to 89.1] | 100.0 [100.0 to 100.0] | 87.5 [38.7 to 98.1] | 77.8 [66.3 to 85.7]

4. Secondary Outcome: Monotherapy Only: Percentage of Participants With Progression-Free Survival at 4 Months
Description: PFS is defined as the time (in months) from the date of first dosing until the date of objective PD (as defined by RECIST version 1.1) or death (by any cause in the absence of progression), whichever occurs earlier. Kaplan-Meier estimates at 4 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 4 months
Population: The Tumor Response-Evaluable Set includes all participants in the full analysis set with at least 1 evaluable postbaseline response assessment using RECIST 1.1. Only participants with data collected at Month 4 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 0 | 3 | 6 | 15 | 3 | 9 | 72
percentage of participants | 73.7 [44.1 to 89.2] |  | 33.3 [0.9 to 77.4] | 33.3 [4.6 to 67.6] | 50.3 [22.6 to 72.8] | 100.0 [100.0 to 100.0] | 62.5 [22.9 to 86.1] | 60.8 [48.5 to 71.0]

5. Secondary Outcome: Monotherapy Only: Percentage of Participants With Progression-Free Survival at 6 Months
Description: PFS is defined as the time (in months) from the date of first dosing until the date of objective PD (as defined by RECIST version 1.1) or death (by any cause in the absence of progression), whichever occurs earlier. Kaplan-Meier estimates at 6 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 6 months
Population: The Tumor Response-Evaluable Set includes all participants in the full analysis set with at least 1 evaluable postbaseline response assessment using RECIST 1.1. Only participants with data collected at Month 6 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 0 | 3 | 6 | 15 | 3 | 9 | 72
percentage of participants | 64.5 [33.6 to 83.8] |  | 33.3 [0.9 to 77.4] | 16.7 [0.8 to 51.7] | 33.5 [10.8 to 58.4] | 66.7 [5.4 to 94.5] | 50.0 [15.2 to 77.5] | 50.3 [38.1 to 61.3]

6. Secondary Outcome: Monotherapy Only: Percentage of Participants With Progression-Free Survival at 8 Months
Description: PFS is defined as the time (in months) from the date of first dosing until the date of objective PD (as defined by RECIST version 1.1) or death (by any cause in the absence of progression), whichever occurs earlier. Kaplan-Meier estimates at 8 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 8 months
Population: The Tumor Response-Evaluable Set includes all participants in the full analysis set with at least 1 evaluable postbaseline response assessment using RECIST 1.1. Only participants with data collected at Month 8 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 0 | 3 | 6 | 15 | 3 | 9 | 72
percentage of participants | 64.5 [33.6 to 83.8] |  | 0.0 [NA to NA] — The 95% confidence internal data was not determined as no participants with PFS at Month 8. | 16.7 [0.8 to 51.7] | 16.8 [2.7 to 41.2] | 66.7 [5.4 to 94.5] | 37.5 [8.7 to 67.4] | 44.2 [32.3 to 55.5]

7. Secondary Outcome: Monotherapy Only: Percentage of Participants With Progression-Free Survival at 10 Months
Description: PFS is defined as the time (in months) from the date of first dosing until the date of objective PD (as defined by RECIST version 1.1) or death (by any cause in the absence of progression), whichever occurs earlier. Kaplan-Meier estimates at 10 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 10 months
Population: The Tumor Response-Evaluable Set includes all participants in the full analysis set with at least 1 evaluable postbaseline response assessment using RECIST 1.1. Only participants with data collected at Month 10 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 0 | 3 | 6 | 15 | 3 | 9 | 72
percentage of participants | 55.2 [25.2 to 77.5] |  | 0.0 [NA to NA] — The 95% confidence internal data was not determined as no participants with PFS at Month 10. | 16.7 [0.8 to 51.7] | 16.8 [2.7 to 41.2] | 0.0 [NA to NA] — The 95% confidence internal data was not determined as no participants with PFS at Month 10. | 12.5 [0.7 to 42.3] | 35.9 [24.6 to 47.3]

8. Secondary Outcome: Monotherapy Only: Percentage of Participants With Progression-Free Survival at 12 Months
Description: PFS is defined as the time (in months) from the date of first dosing until the date of objective PD (as defined by RECIST version 1.1) or death (by any cause in the absence of progression), whichever occurs earlier. Kaplan-Meier estimates at 12 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 12 months
Population: The Tumor Response-Evaluable Set includes all participants in the full analysis set with at least 1 evaluable postbaseline response assessment using RECIST 1.1. Only participants with data collected at Month 12 are reported.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 0 | 3 | 6 | 15 | 3 | 9 | 72
percentage of participants | 27.6 [6.9 to 53.9] |  | 0.0 [NA to NA] — The 95% confidence internal data was not determined as no participants with PFS at Month 12. | 16.7 [0.8 to 51.7] | 16.8 [2.7 to 41.2] | 0.0 [NA to NA] — The 95% confidence internal data was not determined as no participants with PFS at Month 12. | 12.5 [0.7 to 42.3] | 26.2 [15.8 to 37.8]

9. Secondary Outcome: Monotherapy Only: Percentage of Participants With Overall Survival (OS) at 2 Months
Description: OS is defined as the time from the date of enrollment to the date of death from any cause. Kaplan-Meier estimates at 2 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 2 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
percentage of participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 98.7 [90.9 to 99.8]

10. Secondary Outcome: Monotherapy Only: Percentage of Participants With Overall Survival at 4 Months
Description: OS is defined as the time from the date of enrollment to the date of death from any cause. Kaplan-Meier estimates at 4 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 4 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
percentage of participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [47.3 to 98.5] | 97.3 [89.6 to 99.3]

11. Secondary Outcome: Monotherapy Only: Percentage of Participants With Overall Survival at 6 Months
Description: OS is defined as the time from the date of enrollment to the date of death from any cause. Kaplan-Meier estimates at 6 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 6 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
percentage of participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [47.3 to 98.5] | 97.3 [89.6 to 99.3]

12. Secondary Outcome: Monotherapy Only: Percentage of Participants With Overall Survival at 8 Months
Description: OS is defined as the time from the date of enrollment to the date of death from any cause. Kaplan-Meier estimates at 8 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 8 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
percentage of participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [47.3 to 98.5] | 94.0 [84.8 to 97.7]

13. Secondary Outcome: Monotherapy Only: Percentage of Participants With Overall Survival at 10 Months
Description: OS is defined as the time from the date of enrollment to the date of death from any cause. Kaplan-Meier estimates at 10 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 10 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
percentage of participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 83.3 [27.3 to 97.5] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [47.3 to 98.5] | 90.0 [78.8 to 95.4]

14. Secondary Outcome: Monotherapy Only: Percentage of Participants With Overall Survival at 12 Months
Description: OS is defined as the time from the date of enrollment to the date of death from any cause. Kaplan-Meier estimates at 12 months and their confidence intervals are calculated with the log-log transformation methodology of Kalbfleisch and Prentice.
Time Frame: 12 months
Population: as for baseline characteristics
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
percentage of participants | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 83.3 [27.3 to 97.5] | 100.0 [100.0 to 100.0] | 100.0 [100.0 to 100.0] | 90.0 [47.3 to 98.5] | 84.2 [69.8 to 92.1]

15. Secondary Outcome: Objective Response Rate (ORR) for ZN-c5 as a Monotherapy
Description: ORR is defined as the number of participants with measurable disease who have at least 1 confirmed response of CR or PR prior to any evidence of progression (as defined by RECIST v1.1).
Time Frame: 24 weeks
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD
Number analyzed (Participants) | 16 | 3 | 3 | 6 | 15 | 3 | 10 | 75
Participants | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 3

ADVERSE EVENTS:
Time Frame: 12 months
Description: For the safety analysis, Phase 1 Monotherapy group was combined with Phase 2 Monotherapy group.
Arm/Group | Phase 1 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg QD | Phase 1 (Monotherapy): ZN-c5 100 mg QD | Phase 1 (Monotherapy): ZN-c5 75 mg BID | Phase 1 (Monotherapy): ZN-c5 150 mg QD | Phase 1 (Monotherapy): ZN-c5 150 mg BID | Phase 1 (Monotherapy): ZN-c5 300 mg QD | Phase 2 (Monotherapy): ZN-c5 50 mg QD | Phase 1 (Combination Therapy): ZN-c5 25mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 25mg BID + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 50mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 50mg BID + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 100mg QD + Palbociclib | Phase 1 (Combination Therapy): ZN-c5 150mg QD + Palbociclib
All-Cause Mortality (participants affected / at risk) | 4/16 | 1/3 | 1/3 | 2/6 | 6/15 | 1/3 | 4/10 | 8/75 | 2/10 | 3/5 | 2/18 | 0/2 | 4/12 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/3 | 1/3 | 1/6 | 2/15 | 0/3 | 2/10 | 9/75 | 4/10 | 1/5 | 2/18 | 0/2 | 2/12 | 1/3
Other Adverse Events (participants affected / at risk) | 15/16 | 3/3 | 3/3 | 6/6 | 14/15 | 3/3 | 10/10 | 55/75 | 10/10 | 5/5 | 18/18 | 2/2 | 12/12 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Monotherapy): ZN-c5 50 mg QD (N=16) | Phase 1 (Monotherapy): ZN-c5 75 mg QD (N=3) | Phase 1 (Monotherapy): ZN-c5 100 mg QD (N=3) | Phase 1 (Monotherapy): ZN-c5 75 mg BID (N=6) | Phase 1 (Monotherapy): ZN-c5 150 mg QD (N=15) | Phase 1 (Monotherapy): ZN-c5 150 mg BID (N=3) | Phase 1 (Monotherapy): ZN-c5 300 mg QD (N=10) | Phase 2 (Monotherapy): ZN-c5 50 mg QD (N=75) | Phase 1 (Combination Therapy): ZN-c5 25mg QD + Palbociclib (N=10) | Phase 1 (Combination Therapy): ZN-c5 25mg BID + Palbociclib (N=5) | Phase 1 (Combination Therapy): ZN-c5 50mg QD + Palbociclib (N=18) | Phase 1 (Combination Therapy): ZN-c5 50mg BID + Palbociclib (N=2) | Phase 1 (Combination Therapy): ZN-c5 100mg QD + Palbociclib (N=12) | Phase 1 (Combination Therapy): ZN-c5 150mg QD + Palbociclib (N=3)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Calculus urinary (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (Monotherapy): ZN-c5 50 mg QD (N=16) | Phase 1 (Monotherapy): ZN-c5 75 mg QD (N=3) | Phase 1 (Monotherapy): ZN-c5 100 mg QD (N=3) | Phase 1 (Monotherapy): ZN-c5 75 mg BID (N=6) | Phase 1 (Monotherapy): ZN-c5 150 mg QD (N=15) | Phase 1 (Monotherapy): ZN-c5 150 mg BID (N=3) | Phase 1 (Monotherapy): ZN-c5 300 mg QD (N=10) | Phase 2 (Monotherapy): ZN-c5 50 mg QD (N=75) | Phase 1 (Combination Therapy): ZN-c5 25mg QD + Palbociclib (N=10) | Phase 1 (Combination Therapy): ZN-c5 25mg BID + Palbociclib (N=5) | Phase 1 (Combination Therapy): ZN-c5 50mg QD + Palbociclib (N=18) | Phase 1 (Combination Therapy): ZN-c5 50mg BID + Palbociclib (N=2) | Phase 1 (Combination Therapy): ZN-c5 100mg QD + Palbociclib (N=12) | Phase 1 (Combination Therapy): ZN-c5 150mg QD + Palbociclib (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 5 (5) | 5 (5) | 2 (2) | 12 (12) | 1 (1) | 5 (5) | 2 (2)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pericarditis (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Middle ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uveitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Visual field defect (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 7 (7) | 1 (1) | 2 (2) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 4 (4) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Frequent bowel movements (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lip swelling (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 6 (6) | 2 (2) | 4 (4) | 6 (6) | 3 (3) | 3 (3) | 6 (6) | 0 (0) | 4 (4) | 2 (2)
Oesophageal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 7 (7) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Fatigue (General disorders) | 4 (4) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 3 (3) | 6 (6) | 5 (5) | 2 (2) | 10 (10) | 0 (0) | 3 (3) | 2 (2)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Medical device site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (8) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Device related infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vaginal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Eye contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ALT increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 6 (6) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
AST increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 7 (7) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Blood bicarbonate increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood cholesterol increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 6 (6) | 5 (5) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Blood phosphorus increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-reactive protein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Carbohydrate antigen 27.29 increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carcinoembryonic antigen increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GGT increased (Investigations) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 11 (11) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Low density lipoprotein increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3) | 5 (5) | 1 (1) | 6 (6) | 1 (1) | 3 (3) | 2 (2)
Monocyte count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 3 (3) | 14 (14) | 1 (1) | 7 (7) | 3 (3)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 4 (4) | 1 (1)
Platelet count increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour marker increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Weight increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 7 (7) | 3 (3) | 14 (14) | 1 (1) | 11 (11) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 3 (3) | 1 (1) | 5 (5) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 5 (5) | 0 (0) | 3 (3) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (5) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 4 (4) | 0 (0) | 2 (2) | 9 (9) | 0 (0) | 4 (4) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 5 (5) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Muscle fatigue (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Plantar fasciitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Endometrial cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anosmia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Hyperaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Muscle spasticity (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Affect lability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 6 (6) | 1 (1) | 1 (1) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Libido increased (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mania (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Micturition urgency (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast necrosis (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Premature menopause (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulva cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 7 (7) | 2 (2) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mediastinal mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertrichosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Rosacea (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
In the Phase 2 Monotherapy efficacy analysis, efficacy was to be determined by the clinical benefit rate, combining results with similar treatment groups. The Phase 1 Monotherapy group was combined with Phase 2 Monotherapy group. The Phase 2 Combination part of the study was not initiated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In this study, investigators can share findings only after meeting these conditions:

* Study results disclosed publicly by Sponsor or completed at all sites for 2 years
* Investigator informs Sponsor of publication 30 days before submission
* Communication won't include Sponsor's confidential information
* Investigator removes sponsor's confidential information (other than the study results) and agrees to withhold for an additional 60 days in order to obtain patent protection

DOCUMENTS (2):
  • Study Protocol (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/31/NCT03560531/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-17): https://cdn.clinicaltrials.gov/large-docs/31/NCT03560531/SAP_001.pdf